CLINICAL TRIAL: NCT01434173
Title: Risk of Acute Liver Injury in Users of Antimicrobials in the HealthCore Integrated Research Database Population
Brief Title: Risk of Acute Liver Injury in Users of Antimicrobials
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Collaborators: RTI Health Solutions (Other)
Responsible Party: Sponsor
Other Study IDs: 14705
Record Dates: First submitted 2011-07-08; First posted 2011-09-14 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Drug-Induced Liver Injury
Keywords: Liver Diseases; Anti-Bacterial Agents; Fluoroquinolones; Amoxicillin; Amoxicillin-Potassium Clavulanate Combination; Clarithromycin; Doxycycline; Cefuroxime; Case-Control Studies; Retrospective Studies; Cohort Studies; Epidemiologic Research Design; Epidemiologic Studies; HealthCore Integrated Research Database (non-MESH); United States; Human; Insurance Claim Review
MeSH Terms: conditions — Chemical and Drug Induced Liver Injury; Liver Diseases | interventions — Moxifloxacin; Amoxicillin; Clavulanic Acid; Cefuroxime; Clarithromycin; Doxycycline; Levofloxacin; telithromycin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group 1
  Interventions: Drug: Moxifloxacin (Avelox, BAY12-8039)
- Group 2
  Interventions: Drug: Amoxicillin, Amoxicillin plus clavulanic acid, Cefuroxime, Clarithromycin, Doxycycline, Levofloxacin, Telithromycin

INTERVENTIONS:
Drug: Moxifloxacin (Avelox, BAY12-8039) — Eligible patients who are new users of moxifloxacin during the study period. A new user is defined as a person who has a first recorded dispensing of moxifloxacin during the study period and who has not had a previous recorded dispensing for any of the study antimicrobials during the previous 180 days
  Groups: Group 1
Drug: Amoxicillin, Amoxicillin plus clavulanic acid, Cefuroxime, Clarithromycin, Doxycycline, Levofloxacin, Telithromycin — Eligible patients who are new users of one of the other study antimicrobials (amoxicillin, amoxicillin plus clavulanic acid, cefuroxime, clarithromycin, doxycycline, levofloxacin, or telithromycin) during the study period. A new user is defined as a person who has a first recorded dispensing of a study a study antimicrobial during the study period and who has not had a previous recorded dispensing for any of the study antimicrobials during the previous 180 days.
  Groups: Group 2

SUMMARY:
Moxifloxacin is a broad-spectrum antibacterial agent used to treat common community-acquired respiratory tract infections, complicated intra-abdominal infections, and pelvic inflammatory disease. In the clinical development program, moxifloxacin was associated with some hepatic adverse drug reactions. To evaluate further the hepatic safety profile of moxifloxacin, a retrospective cohort study with nested case-control analysis will be conducted to assess the rate of noninfectious acute liver injury among new users of moxifloxacin and of other antimicrobials prescribed for similar indications, including amoxicillin, amoxicillin plus clavulanic acid, cefuroxime, clarithromycin, doxycycline, levofloxacin, and telithromycin.

The study will be implemented in the population included in the HealthCore Integrated Research Database (HIRD). Eligible patients are adults aged 18 years and older with continuous enrollment in the HIRD for at least 6 months before their first claim for a prescription for a study antimicrobial. Follow-up will start at the date of the first prescription until the date of the earliest of the following events: noninfectious acute liver injury, occurrence of an exclusion criterion, end of study period, disenrollment from database, or death. Patients with chronic alcoholism or cirrhosis, infectious hepatitis, HIV/AIDS, or pregnant women will not be included.

DETAILED DESCRIPTION:
Study design is called 'Cohort study with nested case-control analysis"

ELIGIBILITY:
Inclusion Criteria:

* All persons meeting the following criteria during the study period (July 1, 2001, through March 31, 2009) are eligible for study inclusion:
* First insurance claim for a dispensing of one of the study antimicrobials during the study period ("new users")
* Aged 18 years old or older
* Continuous enrollment in the study database for at least 6 months prior to start of follow-up (which is the date of the first claim for any of the study antimicrobials)
* Patient data defined as acceptable for research purposes according to the quality criteria of the HIRD

Exclusion Criteria:

* Pregnant women
* Patients with chronic alcoholism or cirrhosis
* Patients with history of acute and/or chronic infectious hepatitis or HIV/AIDS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The source of study cohort will be the HealthCore Integrated Research DatabaseTM (HIRD) population, which comprises a broad, clinically rich and geographically diverse spectrum of longitudinal claims data from health plans in the United States of America (US)
Sampling Method: Non-Probability Sample
Enrollment: 1299056 (Actual)
Dates: Start 2001-07; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Incidence ratio of noninfectious acute liver injury fulfilling the International Consensus Meeting criteria for drug-induced liver disorders in the study population during periods of treatment with each of the study antimicrobials and nonuse | From the first day of full exposure of a study antimicrobial (day after the date of dispensing) to the end of follow-up (up to 8 years)
Incidence rate ratio of noninfectious acute liver injury fulfilling the International Consensus Meeting criteria for drug-induced liver disorders during treatment with each of the study antimicrobials compared to that during of nonuse | From the first day of full exposure of a study antimicrobial (day after the date of dispensing) to the end of follow-up (up to 8 years)

SECONDARY OUTCOMES:
Incidence rate and incidence rate ratio of noninfectious severe hepatocellular injury as defined by the Hy's Law criteria modified by the FDA Working Group (FDA Working group, 2000; Temple, 2006; Navarro and Senior, 2006) | From the first day of full exposure of a study antimicrobial (day after the date of dispensing) to the end of follow-up (up to 8 years)
Incidence rate and incidence rate ratio of noninfectious acute liver failure, defined as acute liver injury with evidence of coagulation abnormality and any degree of mental alteration (encephalopathy) (Polson and Lee, 2005) | From the first day of full exposure of a study antimicrobial (day after the date of dispensing) to the end of follow-up (up to 8 years)
Cumulative incidence of noninfections acute liver injury, noninfectious severe hepatocellular injury, and noninfectious acute liver failure at weekly intervals after the start of first episode of treatment with each of the study antimicrobials | From the first day of full exposure of a study antimicrobial (day after the date of dispensing) to the end of follow-up (up to 8 years)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Delaware, United States